CLINICAL TRIAL: NCT05360407
Title: The Effect of Mobile Application-based Information About Before and After Surgery on Anxiety, Distress and Quality of Life of Women With Breast Cancer
Brief Title: The Effect of Mobile Application-based Information About Before and After Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Suleyman Demirel University (Other)
Responsible Party: Principal Investigator, Filiz Salman, Principal Investigator, Suleyman Demirel University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: SuleymanDU-SALMAN-F-001
Record Dates: First submitted 2022-04-23; First posted 2022-05-04 (Actual); Last update posted 2022-05-04 (Actual); Status verified 2022-04

CONDITIONS: Breast Cancer
Keywords: breast cancer; mobile application; mobile health; anxiety; distress; quality of life
MeSH Terms: conditions — Breast Neoplasms; Anxiety Disorders | interventions — Postoperative Period

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): The mobile information application was downloaded from the Android market and installed on the patients' phones, and the patients were taught about how to use it. The patients were given a short information brochure on the use of the mobile application. One week after the surgery, the patients were called and reminded about the use of the application. Three weeks after the surgery, data were collected through telephone interviews using the Patient Follow-up Form, Anxiety, Distress and Quality of Life measurement tools, the Patient Information Satisfaction Questionnaire, and the Mobile Application Evaluation Form.
  Interventions: Other: Using mobile information application about before and after surgery
- Control Group (No Intervention): The patients received routine care and training in the clinic, and no additional intervention was applied. Three weeks after the surgery, data were collected through telephone interviews using the Patient Follow-up Form, Anxiety, Distress and Quality of Life measurement tools, and the Patient Information Satisfaction Questionnaire

INTERVENTIONS:
Other: Using mobile information application about before and after surgery — The mobile application had three sections: Information forum (I), Personal forum (notebook and reminder) (II) and Ask the Researcher (messaging) (III). The information forum (Figure 2) is a section that enables patients to access related articles, pictures, and videos. The personal forum is a section that allows patients to create their notes and use the necessary reminders. Ask the researcher section allows patients to communicate with the researcher via messages.
  The participants could download the mobile application with the name "Breast Cancer Surgery Information Guide" from the Google Play Store and install it on their phones. Users who were authenticated by the researcher were able to access the content with an e-mail and password.
  Arms: Intervention Group

SUMMARY:
Aim and hypothesis: This study was conducted to evaluate the effect of mobile information given to women before and after breast cancer surgery on anxiety, distress, and quality of life. E-mobile information given to women before and after breast cancer surgery reduces the level of anxiety (I) and the level of distress (II), and positively affects their quality of life (III).

Methods: This randomized controlled study was conducted between April and August 2021 in the surgical oncology clinic-outpatient clinics of a university hospital. Patients in the intervention group (n=42) used the mobile information application for one month with routine care. Patients in the control group (n=40) received their routine care. Data were collected with data collection forms one week before and three weeks after surgery.

ELIGIBILITY:
Inclusion Criteria:

* Scheduled for elective surgery due to breast cancer,
* Over 18 years old,
* Read and understand Turkish,
* At least primary school graduates,
* Have internet access,
* Have a smartphone with an android operating system suitable for downloading the mobile application.

Exclusion Criteria:

* Diagnosed with active psychiatric disease,
* Using antidepressant medication,
* Vision problems that prevented them from using the mobile application,
* Scheduled for reconstructive surgery using their own tissue

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 82 (Actual)
Dates: Start 2021-04-01 (Actual); Primary Completion 2021-08-30 (Actual); Study Completion 2021-08-30 (Actual)

PRIMARY OUTCOMES:
Change of NCCN Distress Thermometer score at baseline and one month later | The first measurement was collected one week before surgery. The second measurement was collected 3 weeks after surgery.
  This scale was developed by Roth et al. (1998) to measure psycho-social distress in cancer patients. It consists of the visual analog scale that individuals can apply on their own, consists of only one question, and is used to evaluate the stress situations patients have experienced in the last week and a list of problems. There is a thermometer with numbers from 0 to 10 on the scale. On the distress thermometer, a score of 0 indicates that the individual has never experienced distress, and a score of 10 indicates that he or she has experienced distress at the upper limit.

SECONDARY OUTCOMES:
Change of Hospital Anxiety and Depression Scale score at baseline and one month later | The first measurement was collected one week before surgery. The second measurement was collected 3 weeks after surgery.
  The HAD is a self-report scale used to diagnose anxiety and depression in a short time and to determine the risk group in patients with physical illness and/or applying to primary health care services. Only the Anxiety subscale (HAD-A) was used in this study. Anxiety subscale consists of 7 items (1st, 3rd, 5th, 7th, 9th, 11th and 13th questions). Items 1, 3, 5, 11, and 13 show gradually decreasing severity. The score that can be obtained from the HAD-A ranges between 0 and 21 (min.-max.).
Change of FACT-G Quality of Life Scale score at baseline and one month later | The first measurement was collected one week before surgery. The second measurement was collected 3 weeks after surgery.
  Functional Assessment of Cancer Therapy-General (version 4) Quality of Life Scale consists of 4 dimensions; physical well-being (7 items), social/family well-being (7 items), emotional well-being (6 items), and functional well-being (7 items). There are a total of 27 questions on the scale. The scale has a 5-point Likert-type structure and is scored between 0-4. All questions are used to assess the patients' quality of life in the last 7 days. The total score of the scale is equal to the sum of the sub-dimensions, and a high score on the scale indicates a high quality of life.

CONTACTS AND LOCATIONS:
Locations (1):
- Suleyman Demirel University, Isparta, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
Study information will be shared in line with the appropriate requests of researchers via e-mail.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Study information will be shared in line with the appropriate requests of researchers via e-mail.
Access Criteria: Study information will be shared in line with the appropriate requests of researchers via e-mail.

REFERENCES:
- [Background] Barr K, Hill D, Farrelly A, Pitcher M, White V. Unmet information needs predict anxiety in early survivorship in young women with breast cancer. J Cancer Surviv. 2020 Dec;14(6):826-833. doi: 10.1007/s11764-020-00895-7. Epub 2020 Jun 8. PMID 32514909
- [Background] Brennan L, Kessie T, Caulfield B. Patient Experiences of Rehabilitation and the Potential for an mHealth System with Biofeedback After Breast Cancer Surgery: Qualitative Study. JMIR Mhealth Uhealth. 2020 Jul 29;8(7):e19721. doi: 10.2196/19721. PMID 32687476
- [Background] Brett J, Boulton M, Watson E. Development of an e-health app to support women prescribed adjuvant endocrine therapy after treatment for breast cancer. Patient Prefer Adherence. 2018 Dec 11;12:2639-2647. doi: 10.2147/PPA.S187692. eCollection 2018. PMID 30587936
- [Background] Chan RJ, Howell D, Lustberg MB, Mustian K, Koczwara B, Ng CC, Kim Y, Napoles AM, Dixit N, Klemanski D, Ke Y, Toh YL, Fitch MI, Crichton M, Agarawal S, Chan A. Advances and future directions in the use of mobile health in supportive cancer care: proceedings of the 2019 MASCC Annual Meeting symposium. Support Care Cancer. 2020 Sep;28(9):4059-4067. doi: 10.1007/s00520-020-05513-x. Epub 2020 May 14. PMID 32405966
- [Background] Chung IY, Jung M, Park YR, Cho D, Chung H, Min YH, Park HJ, Lee M, Lee SB, Chung S, Son BH, Ahn SH, Lee JW. Exercise Promotion and Distress Reduction Using a Mobile App-Based Community in Breast Cancer Survivors. Front Oncol. 2020 Jan 10;9:1505. doi: 10.3389/fonc.2019.01505. eCollection 2019. PMID 31998651
- [Background] Cinar D, Karadakovan A, Erdogan AP. Effect of mobile phone app-based training on the quality of life for women with breast cancer. Eur J Oncol Nurs. 2021 Jun;52:101960. doi: 10.1016/j.ejon.2021.101960. Epub 2021 Apr 18. PMID 33882446
- [Background] Comez S, Karayurt O. The effect of web-based training on life quality and spousal adjustment for women with breast cancer and their spouses. Eur J Oncol Nurs. 2020 Aug;47:101758. doi: 10.1016/j.ejon.2020.101758. Epub 2020 Apr 9. PMID 32659714
- [Background] Foley NM, O'Connell EP, Lehane EA, Livingstone V, Maher B, Kaimkhani S, Cil T, Relihan N, Bennett MW, Redmond HP, Corrigan MA. PATI: Patient accessed tailored information: A pilot study to evaluate the effect on preoperative breast cancer patients of information delivered via a mobile application. Breast. 2016 Dec;30:54-58. doi: 10.1016/j.breast.2016.08.012. Epub 2016 Sep 6. PMID 27611236
- [Background] Hou IC, Lin HY, Shen SH, Chang KJ, Tai HC, Tsai AJ, Dykes PC. Quality of Life of Women After a First Diagnosis of Breast Cancer Using a Self-Management Support mHealth App in Taiwan: Randomized Controlled Trial. JMIR Mhealth Uhealth. 2020 Mar 4;8(3):e17084. doi: 10.2196/17084. PMID 32130181
- [Background] Korkmaz S, Iyigun E, Tastan S. An Evaluation of the Influence of Web-Based Patient Education on the Anxiety and Life Quality of Patients Who Have Undergone Mammaplasty: a Randomized Controlled Study. J Cancer Educ. 2020 Oct;35(5):912-922. doi: 10.1007/s13187-019-01542-1. PMID 31119709
- [Background] Villarreal-Garza C, Lopez-Martinez EA, Martinez-Cannon BA, Platas A, Castro-Sanchez A, Miaja M, Mohar A, Monroy A, Aguila C, Galvez-Hernandez CL. Medical and information needs among young women with breast cancer in Mexico. Eur J Cancer Care (Engl). 2019 Jul;28(4):e13040. doi: 10.1111/ecc.13040. Epub 2019 Apr 22. PMID 31008546
- [Background] Wysocki WM, Mitus J, Komorowski AL, Karolewski K. Impact of preoperative information on anxiety and disease-related knowledge in women undergoing mastectomy for breast cancer: a randomized clinical trial. Acta Chir Belg. 2012 Mar-Apr;112(2):111-5. doi: 10.1080/00015458.2012.11680807. PMID 22571072